CLINICAL TRIAL: NCT03665675
Title: Pilot Study of Haploidentical or Matched Donor Virus-Specific T-cells (Cytomegalovirus (CMV) or Adenovirus (AdV)) to Treat CMV or AdV Reactivation or Disease in Patients After Solid Organ or Hematopoietic Stem Cell Transplantation (HCT)
Brief Title: Donor Virus-Specific CMV or AdV CTL to Treat CMV or AdV Reactivation or Disease After Solid Organ or HCT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sumithira Vasu (Other)
Responsible Party: Sponsor-Investigator, Sumithira Vasu, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17199; NCI-2018-01412 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-08-13; First posted 2018-09-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation Recipient; Cytomegalovirus; Donor; Solid Organ Transplantation Recipient; Adenovirus
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (CMV-specific CTLs) (Experimental): Participants receive allogeneic cytomegalovirus-specific cytotoxic T lymphocytes IV. Participants with persistent infection are eligible for second infusion after 28 days.
  Interventions: Biological: Allogeneic Cytomegalovirus-Specific Cytotoxic T lymphocytes
- Treatment (AdV-specific CTLs) (Experimental): Patients receive allogeneic adenovirus-specific cytotoxic T Lymphocytes IV. Participants with persistent infection are eligible for second infusion after 28 days.
  Interventions: Biological: Allogeneic Adenovirus-specific Cytotoxic T Lymphocytes

INTERVENTIONS:
Biological: Allogeneic Cytomegalovirus-Specific Cytotoxic T lymphocytes — Given intravenously
  Arms: Treatment (CMV-specific CTLs)
Biological: Allogeneic Adenovirus-specific Cytotoxic T Lymphocytes — Given intravenously
  Arms: Treatment (AdV-specific CTLs)

SUMMARY:
This trial studies the side effects and how well allogeneic cytomegalovirus-specific cytotoxic T lymphocytes (donor cytomegalovirus [CMV] specific cytotoxic T-lymphocytes [CTLs]) or allogeneic adenovirus-specific cytotoxic T lymphocytes (donor adenovirus-specific [AdV] specific CTLs) work in treating CMV or AdV reactivation or infection in participants who have undergone stem cell transplant or solid organ transplant. White blood cells from donors may be able to kill cancer cells in patients with cytomegalovirus or adenovirus that has come back after a stem cell or solid organ transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE I. Assess the safety and feasibility of administering virus specific-CTLs from haploidentical donors in transplant patients both solid organ transplantation (SOT) and hematopoietic cell transplantation (HCT) with CMV/AdV infection despite standard therapy.

OUTLINE:Patients are assigned to 1 of 2 Cohorts.

COHORT A: Patients receive allogeneic cytomegalovirus-specific cytotoxic T lymphocytes intravenously (IV). Patients undergo blood, urine, saliva, cerebrospinal fluid (CSF), and bronchoalveolar fluid sample collection on the trial.

COHORT B: Patients receive allogeneic adenovirus-specific cytotoxic T Lymphocytes IV. Patients undergo blood, urine, saliva, CSF, and bronchoalveolar fluid sample collection on the trial.

After completion of study treatment, participants are followed up at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have solid organ transplant or have received allogeneic hematopoietic stem cell transplant.
* • Cohort A (CMV): Must have documented CMV disease or reactivation, as by:

  * Viremia as detected by quantitative polymerase chain reaction (PCR) (> 500 IU/ml) in the peripheral blood requiring treatment OR
  * High risk for antiviral failure due to history of recurrent CMV reactivations or evidence of antiviral drug resistance, OR
  * Unable to tolerate antiviral drugs due to renal toxicity, bone marrow suppression, transfusion dependent anemia and thrombocytopenia or neutropenia requiring growth factor support or other related organ injury

    • Cohort B (AdV): Must have documented AdV infection or reactivation, as by:
  * Symptomatic subject with any detectable viral load in blood, OR
  * Symptomatic subject with qualitative AdV detection in compartment of current symptomatology, including stool, urine, and/or other specimens (bronchoalveolar lavage (BAL), nasal swab, CSF, etc.), irrespective of blood viral load, OR
  * New, persistent, and/or worsening AdV-related symptoms, signs, and/or markers of end organ compromise while receiving antiviral therapy (ie cidofovir), OR
  * Asymptomatic with a viral load > 1000 copies/ml in peripheral blood, OR
  * Unable to tolerate antiviral treatment due to renal toxicity, bone marrow suppression, transfusion dependent anemia and thrombocytopenia or neutropenia requiring growth factor support or other related organ injury

    * Karnofsky (age > 16 years) or Lansky performance score > 70 (age < 16)
    * Available seropositive haploidentical or matched donor who is without evidence of infection that would otherwise preclude donation
    * Negative pregnancy test in female patients if applicable (childbearing potential, has not received a full-intensity conditioning regimen
    * Written informed consent and/or signed assent line from patient, parent or guardian
    * DONOR
    * Human leukocyte antigen (HLA)-haploidentical or full-match to the patient as determined by institutional standards
    * Cohort A: CMV seropositive, defined as detection of serum CMV immunoglobulin G (IgG)
    * Cohort B: AdV seropositive, defined as detection of serum AdV IgG
    * Age 18 or over
    * Meet donor eligibility or suitability according to institutional standards. If the donor is deemed ineligible according to Foundation for the Accreditation of Cellular Therapy (FACT) standards, but is suitable for donation per institutional standards, the donor will be eligible for the protocol

Exclusion Criteria:

* Receipt of anti-thymocyte globulin (ATG), alemtuzumab, or other T-cell depleting agents within 21 days of screening for enrollment.
* Receipt of > 0.5mg/kg/day of prednisone or steroid equivalent at the time of enrollment. Stable GVHD is permitted as long as patients are on stable dose steroids of less than or equal to 0.5 mg/kg/day of prednisone or steroid equivalent.
* Evidence of uncontrolled infection as follows:

  * Bacterial infections - patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment.
  * Fungal infections - patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment.
  * Patients with hemodynamic instability attributable to bacterial sepsis or new symptoms, worsening physical signs or radiographic findings attributable to concomitant bacterial or fungal infection are excluded. Patients who require ventilator support for CMV pneumonitis are not excluded. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Receipt of donor lymphocyte infusion (DLI) within 28 days.
* Patients with active acute graft versus host disease (GvHD) grades II-IV requiring > 0.5 mg/kg/day of prednisone or steroid equivalent or T-cell depleting immunosuppression.
* Acute graft rejection in solid organ transplantation requiring augmented immunosuppression with T-cell depleting agents or steroids as mentioned above.
* Active and uncontrolled relapse of malignancy.

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-07 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events defined by the National Cancer Institute Common Terminology Criteria for Adverse Events 4.0 | Up to 30 days post infusion
  Measured as the proportion of patients with acute (a) graft versus host disease (GvHD) grades III-IV or graft rejection/failure within 30 days of the last dose of cytotoxic T-lymphocytes (CTLs) or grades 3-5 infusion-related adverse events within 7 days of the last does of CTLs or grades 4-5 non-hematological adverse events within 30 days of the last dose of CTLs and that are not due to the pre-existing infection or the original malignancy or pre-existing co-morbidities. Will be calculated by dividing by all evaluable patients and the corresponding 95% confidence intervals will be calculated.
Feasibility defined as identifying a suitable donor within 4 weeks and meeting minimum T cell doses in the final product | Up to 1 year

SECONDARY OUTCOMES:
Antiviral activity defined as response to viral load | At day 28
  Complete response, partial response, stable disease or progression will be defined and proportion of each outcome will be calculated.
Persistence of infused CTLs as measured by T cell gene rearrangement and effects on clinical signs of viral infection | Up to 1 year
Overall survival | From last CTL infusion till death, assessed at 6 and 12 months
  Kaplan-Meier survival function will be used to estimate the survival probability.
Risk for chronic GVHD | At 6 and 12 months post CTL infusion
  Survival analysis method will be applied. Time to chronic GVHD will be defined from time of the last CTL infusion to the onset of chronic GVHD, or the last clinical assessment date if no chronic GVHD. Cumulative incidence of chronic GVHD at 6 and 12 months will be estimated.
Systemic infections | Within 6 months of CTL infusion
  Will be reported by etiologic agent, site of disease, date of onset, and severity.
Secondary graft failure | 30 days post-CTL infusion
  Proportion of secondary graft failure for both populations will be assessed at 30 days post CTL infusion will be calculated and 95% confidence intervals will be estimated accordingly.
Effects of cytomegalovirus (CMV) specific-CTL on viral loads assessed by weekly reverse transcriptase-polymerase chain reaction | Up to 1 year
Viral reactivations | Up to 6 months
  Proportion of viral reactivations within 6 months will be calculated and 95% confidence intervals will be estimated accordingly.
Clinical response to CTL infusions | At 6 weeks and 3 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0". | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sumithira Vasu, MBBS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu